CLINICAL TRIAL: NCT03876873
Title: A Prospective, Randomized, Non-Blinded, Crossover Controlled Clinical Trial Evaluating the Efficacy of Face Mask Ventilation With 45 Degree Head Rotation in Anesthetized Obese (BMI ≥ 35) Adults
Brief Title: Effect of Head Rotation on Efficacy of Face Mask Ventilation in Anesthetized Obese (BMI ≥ 35) Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Boris Mraovic, Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2012364
Record Dates: First submitted 2019-03-13; First posted 2019-03-15 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Noninvasive Ventilation
Keywords: Face Mask; Obesity; Anesthetized Adult; Ventilation; Head Rotation
MeSH Terms: conditions — Obesity; Respiratory Aspiration | interventions — Masks

STUDY DESIGN:
Intervention Model Description: Participants will be assigned into one of two groups (per a randomization schedule) for face mask ventilation. The sequence of face mask ventilation head positions will be determined by group assignment. Each position will be performed for one minute. Group A: (1) neutral position, (2) head rotation, (3) neutral position. Group B: (1) head rotation, (2) neutral position, (3) head rotation.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The surgeon, anesthesiologist, operating room staff, and participants will not know the group assignment at the time of subject recruitment. No blinding will occur during the clinical portion of the study or during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Group A (Experimental): Head Rotation During Face Mask Ventilation. Step 1: Neutral Position (1 minute), Step 2: Head Rotation (1 minute), Step 3: Neutral Position (1 minute)
  Interventions: Procedure: Head Rotation During Face Mask Ventilation; Device: Medline Top Valve Anesthesia Mask
- Group B (Experimental): Head Rotation During Face Mask Ventilation. Step 1: Head Rotation (1 Minute), Step 2: Neutral Position (1 minute), Step 3, Head Rotation (1 Minute)
  Interventions: Procedure: Head Rotation During Face Mask Ventilation; Device: Medline Top Valve Anesthesia Mask

INTERVENTIONS:
Procedure: Head Rotation During Face Mask Ventilation — Participants will receive face mask ventilation in either a neutral head position (practice standard position) or a head rotation position (45 degree angle).
Device: Medline Top Valve Anesthesia Mask — Face mask used per standard of care to provide oxygen to subjects before surgical procedures.
  Other Names: Face Mask

SUMMARY:
Mask ventilation is fundamental to airway management at the start of surgical procedures requiring general anesthesia. For general anesthesia, medications are provided that affect the entire body and lead to a loss of consciousness. Medical professionals perform mask ventilation by placing a plastic mask over a subjects mouth and nose to provide enough oxygen for the placement of a breathing tube. In this study, we expect that a 45 degree rotation of the head will increase the efficiency of mask ventilation.

DETAILED DESCRIPTION:
Mask ventilation is a foundation of airway management after the initial induction of anesthesia. It allows for adequate oxygenation of the patient to buy enough time for intubation, during which the patient is not ventilated. However, in some patients mask ventilation may be difficult - older than 55 years, heavier (BMI > 26 kg/m^2), with no teeth, having a beard or sleep apnea. Inadequate ventilation, if not corrected, can result in decreasing oxygen saturation to dangerous levels - which could lead to devastating complications. As a result, the efficacy of mask ventilation is of critical importance to patient safety after the induction of anesthesia.

A recent study proposed that mask ventilation could be improved simply by turning a patient's head. The study showed that rotating a patient's head to a 45 degree angle significantly improved mask ventilation when compared with the head placed in a neutral position. However, this study was done in patients with a BMI lass than 35. As such, the effects of head rotation on the efficacy of mask ventilation has not been studied in patients with a BMI of 35 and greater.

Obesity (BMI ≥ 30 kg/m^2) affects almost 40% of US adults and is one of the most prevalent health concerns in our society. It is a predictor of difficult mask ventilation because it is associated with increased upper airway obstruction, decreased airway patency, and decreased lung volumes such as functional residual capacity (FRC). If previous findings in regard to the effects of 45 degree head rotation on the efficacy of ventilation hold true in the obese patient, then this study will show that head rotation could be used as a simple way to improve the efficacy of mask ventilation for patients with a BMI of 35 and above.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ASA Physical Status Classification I-III
* Body Mass Index (BMI) ≥ 35 kg/m^2

Exclusion Criteria:

* Inability to obtain written informed consent
* Pregnant or breastfeeding
* Limited head rotation or neck extension
* Subjects with expected or history difficult intubation
* Large beard
* Orogastric (OG)/nasogastric (NG) tube
* Gastroesophageal Reflux Disease (GERD)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Mraovic, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langeron O, Birenbaum A, Le Sache F, Raux M. Airway management in obese patient. Minerva Anestesiol. 2014 Mar;80(3):382-92. Epub 2013 Oct 14. PMID 24122033
- [Background] Kheterpal S, Han R, Tremper KK, Shanks A, Tait AR, O'Reilly M, Ludwig TA. Incidence and predictors of difficult and impossible mask ventilation. Anesthesiology. 2006 Nov;105(5):885-91. doi: 10.1097/00000542-200611000-00007. PMID 17065880
- [Background] Kheterpal S, Martin L, Shanks AM, Tremper KK. Prediction and outcomes of impossible mask ventilation: a review of 50,000 anesthetics. Anesthesiology. 2009 Apr;110(4):891-7. doi: 10.1097/ALN.0b013e31819b5b87. PMID 19293691
- [Background] Itagaki T, Oto J, Burns SM, Jiang Y, Kacmarek RM, Mountjoy JR. The effect of head rotation on efficiency of face mask ventilation in anaesthetised apnoeic adults: A randomised, crossover study. Eur J Anaesthesiol. 2017 Jul;34(7):432-440. doi: 10.1097/EJA.0000000000000582. PMID 28009638
- [Background] Hales CM, Carroll MD, Fryar CD, Ogden CL. Prevalence of Obesity Among Adults and Youth: United States, 2015-2016. NCHS Data Brief. 2017 Oct;(288):1-8. PMID 29155689

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A | Group B
Started | 9 | 12
Completed | 9 | 11
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 9 | 12 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 11 | 20
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 17
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 12 | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximal and Average Expiratory Tidal Volume During Mask Ventilation
Description: Measured in mL
Time Frame: Day 1
Population: Both groups' patients' heads were rotated, however, in the Neutral Position group the patients' heads started in neutral position, while the Head Rotation group's heads started in rotated position. Data were not collected for each 1-minute change within the groups.
Measure: Mean (Standard Deviation); unit: Milliliter
Groups:
- Neutral Position: Head Rotation During Face Mask Ventilation. Step 1: Neutral Position (1 minute), Step 2: Head Rotation (1 minute), Step 3: Neutral Position (1 minute) Patients' heads started in neutral position, and was rotated 45 degrees for 1 minute, then returned to neutral position during the 3-minute preoxygenation prior to anesthesia induction.
- Head Rotation: Head Rotation During Face Mask Ventilation. Step 1: Head Rotation (1 Minute), Step 2: Neutral Position (1 minute), Step 3, Head Rotation (1 Minute)
  Patients' heads started in 45 degree rotated position, and was returned to normal position for 1 minute, then returned to 45 degree rotated position during the 3-minute preoxygenation prior to anesthesia induction.
Arm/Group | Neutral Position | Head Rotation
Number analyzed (Participants) | 9 | 11
Milliliter
  Maximal expiratory tidal volume | 25 (11.39) | 26.52 (10.31)
  Average expiratory tidal volume | 21.96 (11.40) | 23.33 (9.90)

2. Secondary Outcome: Maximal and Average Inspiratory Tidal Volume During Mask Ventilation
Description: Measured in mL
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Milliliter
Arm/Group | Neutral Position | Head Rotation
Number analyzed (Participants) | 9 | 11
Milliliter
  Maximal inspiratory tidal volume | 415.48 (182.27) | 395.35 (158.73)
  Average inspiratory tidal volume | 339.86 (243.76) | 296.45 (90.86)

3. Secondary Outcome: Maximal and Average End-tidal CO2 (ETCO2) During Mask Ventilation
Description: Measured in mm Hg
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Neutral Position | Head Rotation
Number analyzed (Participants) | 9 | 11
Millimeters of mercury
  Maximal end-tidal CO2 | 23 (13.88) | 31.36 (5.26)
  Average end-tidal CO2 | 18.59 (12.19) | 23.93 (6.41)

4. Secondary Outcome: Maximal and Average Airway Flow During Mask Ventilation
Description: Measured in L/min
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters per minute
Arm/Group | Neutral Position | Head Rotation
Number analyzed (Participants) | 9 | 11
Liters per minute
  Maximal airway flow | 97.69 (3.21) | 98.03 (2.50)
  Average airway flow | 97.95 (3.90) | 96.78 (3.53)

5. Secondary Outcome: Lowest and Delta O2 Saturation Drop on SpO2 During Mask Ventilation
Description: Measured in %
  Delta O2 saturation drop is the difference between 100% oxygen saturation and the lowest oxygen saturation measured, e.g., 100 - 96 (lowest measured) = 4 (delta).
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Neutral Position | Head Rotation
Number analyzed (Participants) | 9 | 11
Percentage
  Lowest O2 saturation drop on SpO2 | 96.78 (3.53) | 95.73 (3.95)
  Delta O2 saturation drop on SpO2 | 3.22 (3.53) | 4.18 (4.02)

6. Secondary Outcome: Lowest and Delta O2 Saturation Drop on SpO2 During Intubation
Description: as for outcome 5
Time Frame: Day 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Neutral Position | Head Rotation
Number analyzed (Participants) | 9 | 11
Percentage
  Lowest O2 saturation drop on SpO2 | 2.28 (3.22) | 1.90 (2.51)
  Delta O2 saturation drop on SpO2 | 3.22 (3.53) | 4.18 (4.02)

ADVERSE EVENTS:
Time Frame: One day
Description: 1 patient from group B experienced apnea after intubation had been completed.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/12
Other Adverse Events (participants affected / at risk) | 0/9 | 1/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=9) | Group B (N=12)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-24): https://cdn.clinicaltrials.gov/large-docs/73/NCT03876873/Prot_SAP_000.pdf